CLINICAL TRIAL: NCT02238990
Title: Biomarkerscreening Via Transcriptome and Methylosome Analysis in Cervical Cancer and Its Preinvasive Lesions
Brief Title: Biomarkerscreening in Cervical Cancer and Its Preinvasive Lesions
Status: Active, not recruiting | Type: Observational
Sponsor: University of Luebeck (Other)
Responsible Party: Principal Investigator, Daniel Alexander Beyer, Priv.-Doz.Dr.med.habil., University of Luebeck
Other Study IDs: UKSH-HL-14-099; UKSH-HL-14-099 (Other: Ethicscomittee Luebeck 14-099)
Record Dates: First submitted 2014-09-04; First posted 2014-09-12 (Estimated); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Evaluation of New Tissue Biomarkers for Cervical Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — tissue samples of the cervix uteri
Oversight: Data Monitoring Committee: No

SUMMARY:
The following trial is a multicenter and prospective research trial of the colposcopy unit of luebeck university and the national research center in Borstel, Germany.

The study is to identify and evaluate new biomarkers in human papilloma virus (HPV) associated malignancies and its preinvasive lesions of the cervix uteri. Fresh tissue samples being removed during conizations and/or hysterectomies are to be fixed in HOPE's solution and analyzed according to their transcriptomes and methylosome. The hereby found candidates are to be validated using immunohistochemistry and RT [real-time] -PCR [polymerase chain reaction].

The project is meant to be followed by continuous studies developing a new test describing the malignant potential of HPV associated genital lesions.

ELIGIBILITY:
Inclusion Criteria:

* Positive informed consent
* Patients with suspected preinvasive genital lesion
* Patients with confirmed genital lesion (both preinvasive and invasive)
* Contact via dept. of obs/gyn of luebeck university
* Complete set of data

Exclusion Criteria:

* Incomplete set of data
* Negative informed consent

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The population is to be recruted from A. patients suffering from cervical cancer B. patients suffering from preinvasive cervical lesions
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-09 (Actual); Primary Completion 2030-12-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
CIN III (cervical intraepithelial neoplasia) lesions | three years
  number of CIN III lesions
cervical cancer | three years
  number of cervical cancer probes
HPV | three years
  number and type of HPV infection of the analyzed probes

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Beyer, PD Dr., Principal Investigator — University of Luebeck; Torsten Goldmann, Prof. Dr., Principal Investigator — Forschungszentrum Borstel
Locations (1):
- Luebeck University, Department for obstetrics and gynecology, Lübeck, Schleswig-Holstein, Germany

REFERENCES:
- [Background] Apgar BS, Kittendorf AL, Bettcher CM, Wong J, Kaufman AJ. Update on ASCCP consensus guidelines for abnormal cervical screening tests and cervical histology. Am Fam Physician. 2009 Jul 15;80(2):147-55. PMID 19621855
- [Background] Gagne HM. Colposcopy of the vagina and vulva. Obstet Gynecol Clin North Am. 2008 Dec;35(4):659-69; x. doi: 10.1016/j.ogc.2008.10.002. PMID 19061824
- [Background] Massad LS, Jeronimo J, Katki HA, Schiffman M; National Institutes of Health/American Society for Colposcopy and Cervical Pathology Research Group. The accuracy of colposcopic grading for detection of high-grade cervical intraepithelial neoplasia. J Low Genit Tract Dis. 2009 Jul;13(3):137-44. doi: 10.1097/LGT.0b013e31819308d4. PMID 19550210